CLINICAL TRIAL: NCT06905314
Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HRS-4029 Following a Single Dose in Healthy Subjects
Brief Title: A Single Ascending Dose of HRS-4029 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-4029-101
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): Drug: HRS-4029 Subject will receive HRS-4029 at dose level 1. Drug: Placebo Subject will receive placebo at dose level 1.
  Interventions: Drug: HRS-4029; Drug: Placebo
- Group B (Experimental): Drug: HRS-4029 Subject will receive HRS-4029 at dose level 2. Drug: Placebo Subject will receive placebo at dose level 2.
  Interventions: Drug: HRS-4029; Drug: Placebo
- Group C (Experimental): Drug: HRS-4029 Subject will receive HRS-4029 at dose level 3. Drug: Placebo Subject will receive placebo at dose level 3.
  Interventions: Drug: HRS-4029; Drug: Placebo
- Group D (Experimental): Drug: HRS-4029 Subject will receive HRS-4029 at dose level 4. Drug: Placebo Subject will receive placebo at dose level 4.
  Interventions: Drug: HRS-4029; Drug: Placebo
- Group E (Experimental): Drug: HRS-4029 Subject will receive HRS-4029 at dose level 5. Drug: Placebo Subject will receive placebo at dose level 5.
  Interventions: Drug: HRS-4029; Drug: Placebo
- Group F (Experimental): Drug: HRS-4029 Subject will receive HRS-4029 at dose level 6. Drug: Placebo Subject will receive placebo at dose level 6.
  Interventions: Drug: HRS-4029; Drug: Placebo

INTERVENTIONS:
Drug: HRS-4029 — HRS-4029
Drug: Placebo — Placebo

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and pharmacokinetics of HRS-4029 following a single intravenous dose administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 55 years.
2. Body mass index (BMI) of 19.0 to 28.0 kg/m2 (inclusive).
3. Agreed to take effective contraceptive measures during and 3 months after the last dose of the study period.
4. Understand in detail the content, procedure and possible adverse effects of the trial, and voluntarily sign the written informed consent form (ICF).

Exclusion Criteria:

1. Diseases with abnormal clinical manifestations that occurred before screening or are currently occurring and need to be excluded.
2. Vital signs, physical examination, 12-lead electrocardiogram,or laboratory examination deemed clinically significant by the investigator .
3. Subjects with positive tests for infectious diseases.
4. Female who are pregnant or breastfeeding.
5. Unable to tolerate venipunctures or have a history of fainting needles and blood.
6. Historic abuse of alcoholic beverages
7. Smoke ≥5 cigarettes per day within 3 months prior to the study
8. History of drug abuse.
9. Other reasons that the investigator consider it inappropriate to participate in the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | From ICF signing date to Day15

SECONDARY OUTCOMES:
Maximum observed concentration of HRS-4029 (Cmax) | 0 hour to 48 hour after administration
Area under the serum concentration time curve (AUC) of HRS-4029 | 0 hour to 48 hour after administration
Time to maximum observed concentration (Tmax) of HRS-4029 | 0 hour to 48 hour after administration
Half-life (T1/2) of HRS-4029 | 0 hour to 48 hour after administration
Clearance (CL) of HRS-4029 | 0 hour to 48 hour after administration
Volume of distribution (Vz) of HRS-4029 | 0 hour to 48 hour after administration
Number of subjects who developed HRS-4029 antidrug antibodies (ADA) | Baseline to Day15

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided